CLINICAL TRIAL: NCT07075744
Title: Association Between Intraoperative Heart Rate and Postoperative 30-day Mortality in Non-cardiac Surgery
Brief Title: Intraoperative Heart Rate Thresholds and Postoperative Mortality
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sung-Hoon Kim, Associate Professor, Asan Medical Center
Other Study IDs: AMC [2023-0611]
Record Dates: First submitted 2025-07-11; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: HEART RATE
Keywords: Heart rate; Intraoperative; Tachycardia; Bradycardia; Mortality
MeSH Terms: conditions — Tachycardia; Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Non-cardiac Surgery Cohort: This cohort includes adult patients who underwent non-cardiac surgery under general or regional anesthesia. The study retrospectively examined intraoperative heart rate patterns and their association with postoperative 30-day mortality. No intervention was applied as this is an observational study.
  Interventions: Other: Intraoperative Heart Rate Monitoring

INTERVENTIONS:
Other: Intraoperative Heart Rate Monitoring — This is a non-interventional observational analysis of intraoperative heart rate metrics, including minimum, maximum, average, and time-weighted average heart rate recorded during non-cardiac surgery. The study also includes duration-based metrics such as time spent below or above specific heart rate thresholds. These variables were retrospectively analyzed for their association with 30-day postoperative mortality. No clinical intervention or treatment was administered as part of this study.

SUMMARY:
This retrospective observational study investigates the association between intraoperative heart rate and 30-day postoperative mortality among patients undergoing non-cardiac surgery. The findings suggest that heart rate abnormalities during surgery may significantly affect short-term postoperative outcomes.

DETAILED DESCRIPTION:
This is a retrospective cohort study conducted to evaluate the clinical impact of intraoperative heart rate on postoperative 30-day mortality in patients undergoing non-cardiac surgery. Patient data were extracted from a large institutional electronic medical record database, including demographic variables, comorbidities, anesthesia records, and perioperative outcomes.

Heart rate was continuously recorded at 1-minute or 5-minute intervals during the surgery. Various heart rate parameters-such as minimum, maximum, average, and time-weighted average-were analyzed, and threshold-based metrics (e.g., minutes spent below or above defined thresholds) were computed using a piecewise cubic Hermite interpolating polynomial (PCHIP) method to smooth minute-by-minute fluctuations.

The primary outcome was all-cause mortality within 30 days after surgery. Multivariable logistic regression and sensitivity analyses were performed to adjust for potential confounders. The study aimed to provide clinical insight into the prognostic value of intraoperative heart rate dynamics and to identify modifiable intraoperative risk factors for mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent non-cardiac surgery at our medical center between March 2019 and February 2023
* Age ≥ 18 years
* Availability of complete laboratory data and perioperative vital signs
* Only the first surgery performed after hospital admission was included for patients with multiple

Exclusion Criteria:

* Cardiac-related surgical procedures
* Pregnancy at the time of surgery
* Age < 18 years
* Surgeries lasting less than 30 minutes
* Cadaveric procedures
* Missing or incomplete laboratory values or vital sign data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients (aged 18 years or older) who underwent non-cardiac surgery under general or regional anesthesia at a single tertiary medical center. Only the first surgery after admission was included for patients who underwent multiple procedures. Patients undergoing cardiac-related procedures, pediatric or obstetric cases, cadaveric surgeries, or those with incomplete vital signs or laboratory data were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 139149 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
All-cause mortality within 30 days after non-cardiac surgery | 30 days after the date of surgery
  The primary outcome is defined as death from any cause occurring within 30 days after the date of surgery. Mortality data were collected from institutional electronic medical records and verified through discharge and follow-up records. The association between intraoperative heart rate metrics and postoperative mortality was retrospectively analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: No
The dataset used and/or analyzed during the current study is available from the corresponding author upon reasonable request.